CLINICAL TRIAL: NCT05283603
Title: Registro Osservazionale Dei Pazienti Con Blocco Della Branca Sinistra
Brief Title: Clinical Observational Registry of Patients With Left Bundle Branch Block
Acronym: RECOrd-LBBB
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria di Sassari (Other)
Responsible Party: Principal Investigator, Giuseppe Damiano Sanna, MD PhD, Azienda Ospedaliero Universitaria di Sassari
Other Study IDs: PG/2019/8862
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Left Bundle Branch Block (LBBB) on ECG
MeSH Terms: conditions — Bundle-Branch Block | interventions — Electrocardiography; Echocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG, Echocardiogram, Magnetic resonance — Clinical and instrumental follow-up

SUMMARY:
The electromechanical dyssynchrony induced by the presence of LBBB is in some patients, but not all, the cause of progressive left ventricular systolic dysfunction and heart failure.

Aims

1. To investigate the clinical, ECG, imaging-derived features in a large cohort of patients affected by LBBB on ECG.
2. To identify predictors of LBBB-induced LV systolic dysfunction and predictors of outcome in this population.
3. To derive data which may have an impact on therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* LBBB on ECG

Exclusion Criteria:

* Previous extensive anterior myocardial infarction
* Previous cardiac surgery or transcatheter aortic valve implantation (TAVI)
* Congenital structural heart disease
* Patients implanted with permanent right ventricular stimulation devices and permanent pacing
* Denial to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with LBBB
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular dysfunction | 20 years
  Echocardiographic left ventricular ejection fraction - EF (%)

SECONDARY OUTCOMES:
Adverse cardiovascular events (e.g., heart failure) | 20 years
  Heart failure (incidence and prevalence) Hospitalizations due to heart failure MACE

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology, AOU Sassari, Sassari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanna GD, De Bellis A, Zecchin M, Beccu E, Carta P, Moccia E, Canonico ME, Parodi G, Sinagra G, Merlo M. Prevalence, clinical and instrumental features of left bundle branch block-induced cardiomyopathy: the CLIMB registry. ESC Heart Fail. 2021 Dec;8(6):5589-5593. doi: 10.1002/ehf2.13568. Epub 2021 Sep 12. PMID 34510787
- [Background] Sanna GD, Merlo M, Moccia E, Fabris E, Masia SL, Finocchiaro G, Parodi G, Sinagra G. Left bundle branch block-induced cardiomyopathy: a diagnostic proposal for a poorly explored pathological entity. Int J Cardiol. 2020 Jan 15;299:199-205. doi: 10.1016/j.ijcard.2019.06.008. Epub 2019 Jun 4. PMID 31186131
- [Background] Moccia E, Sanna GD, Parodi G. Transient left bundle branch block and intraventricular dyssynchrony as a cause of reversible left ventricular dysfunction: The "in vivo" documentation of spontaneous electrical remodeling. Ann Noninvasive Electrocardiol. 2019 Nov;24(6):e12667. doi: 10.1111/anec.12667. Epub 2019 May 29. PMID 31141243